CLINICAL TRIAL: NCT06609681
Title: Flipping the Paradigm of Parkinson Disease: A Model of National Eat, Move, Sleep Digital Interventions to Prevent or Slow a Rise of Non-Communicable Diseases in Thailand
Brief Title: Parkinson Disease: A Model of National Digital Interventions to Prevent or Slow a Rise of Non-Communicable
Acronym: PDRegistry
Status: Active, not recruiting | Type: Observational
Sponsor: Roongrooj Bhidayasiri (Other)
Responsible Party: Sponsor-Investigator, Roongrooj Bhidayasiri, Chulalongkorn Center of Excellence for Parkinson is disease and related to movement disorder, Chulalongkorn Centre of Excellence for Parkinson's Disease and Related Disorders
Organization: Chulalongkorn Centre of Excellence for Parkinson's Disease and Related Disorders (Other)
Other Study IDs: Med Chula IRB No.0804/65; GCE 3300160003 (Other: Center of Excellence grant of Chulalongkorn, Thailand.)
Record Dates: First submitted 2024-09-16; First posted 2024-09-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Thai Parkinson Screening. Registry.
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to Parkinson's Disease Medical Center of Excellence's project which was registered Parkinson's disease patients in 2008-2011, it was found that there were more than 60,000 people with Parkinson's disease in Thailand, approximately 1 over 3 of all elderly people.

It is estimated that the prevalence of Parkinson's disease is approximately 242.57 per 100,000 people of all elderly people, and it is likely to increase due to the current situation of Thailand which is entering aging society. The current diagnosis of Parkinson's disease still relies heavily on medical history and physical examination. The accuracy of diagnosing Parkinson's disease by neurologists is approximately 80 percent, especially when they have been following up consistently. Nonetheless, if they have Parkinson's disease in the early stages, the signs and symptoms will not be severe. Therefore, diagnostic accuracy will decrease around 40-50 percent, making it difficult to diagnose Parkinson's disease patients at an early stage and as a consequence, there still are many undiagnosed patients in 2022. Consequently, Parkinson's Disease Medical Center of Excellence is planning to establish this pilot research project to develop and analyze advanced data of the screening system for people at risk and precursor symptoms to Parkinson's disease, Chulalongkorn Hospital, Thai Red Cross Society. Dividing patients into 3 groups, those who have precursor symptoms, who are at risk of developing disease and Parkinson's disease patients, using the digital platform on mobile application that includes general information, health information, congenital diseases, regularly used medications, initial abnormal symptoms, various risk factors, writing and handwriting, pronunciation assessments, and get diagnosis from experts for referral in the public health system.

DETAILED DESCRIPTION:
1. Flipping the Paradigm of Parkinson's Disease: A Model of National 'Eat, Move, Sleep' Digital Interventions to Prevent or Slow a Rise of Non-Communicable Diseases in Thailand
2. Principal Investigator: Roongroj Bhidayasiri
3. Study centers and Address: Chulalongkorn Center of Excellence for Parkinson's disease and related to movement disorder 1183 RAMA 4 Rd. Pathum wan, Bangkok 10330 and 76 provinces of Thailand.

The Screening of Parkinson's patients with digital technology and sensors and analyze with artificial intelligence the following information

1. Innovative prototype questionnaire. Screening of Parkinson's patients with digital technology.
2. Sound screening that can detect speech
3. Handwriting test by writing sentences and spiral circles.
4. Testing finger dexterity and alternating tap test
5. Tremor analysis
6. Gait analysis
7. Assessing your ability to get out of bed
8. Sleep quality
9. Sleep assessment by polysomnography test
10. Ability to smell

ELIGIBILITY:
Inclusion Criteria:

1. Thai Adult age more than 40 years old.
2. Family history with Parkinson's disease.

Exclusion Criteria:

1. Thai Adult age less than 40 years old

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Thai Adult age more than 40year old
Study Population: - Thai Adult age more than 40year old or have family history of Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Digital platform system; Motor and non-motor symptom of Parkinson' s disease questionnaire, tremor and voice test | 1 year
  a web-based structural software package that speeds and eases transactions among users. Digital platforms serve digital markets, while also offering physical products.

SECONDARY OUTCOMES:
Age | 1 year
  the number of years that someone has lived, or that something has existed
Early Lifestyle interventions Eat Move Sleep | 1 year
  Early detection, especially for early PD, prodromal PD, and individuals at risk for PD.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Roongroj Bhidayasiri, M.D., Principal Investigator — Chulalongkorn Centre of Excellence for Parkinson's Disease and Related Disorders
Locations (1):
- Chulalongkorn Center of Excellence for Parkinson's disease and related to movement disorder, Pathum Wan, Bangkok, Thailand

DOCUMENTS (1):
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT06609681/ICF_000.pdf